CLINICAL TRIAL: NCT04789603
Title: Effects of Using the Surgical Mask and FFp2 in the Distance Walked, Heart Rate, Oxygenometry, and Tone of the Accessory Inspiratory Muscles During the 6-minute Walking Test
Brief Title: Effects of Using Mask During the 6-minute Walking Test in Times of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez Sanz, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: CBAS-2020-03
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Disease; Covid19; Physical Disability
Keywords: covid-19; muscle tone; mask
MeSH Terms: conditions — Lung Diseases; COVID-19 | interventions — Walking; Masks

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: For randomization a computer software (www.random.org) will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Without Mask Group (Active Comparator): Patients who will perform the 6-min walk test without mask
  Interventions: Other: 6-min-walk without mask
- Surgical Mask (Active Comparator): Patients who will perform the 6-min walk test with surgical mask
  Interventions: Other: 6-min-walk surgical mask
- Fpp2 Mask (Experimental): Patients who will perform the 6-min walk test with Fpp2 mask
  Interventions: Other: 6-min-walk Fpp2

INTERVENTIONS:
Other: 6-min-walk surgical mask — To walk as fast as possible without running for 6 minutes with surgical mask
  Arms: Surgical Mask
Other: 6-min-walk Fpp2 — To walk as fast as possible without running for 6 minutes with Fpp2 mask
  Arms: Fpp2 Mask
Other: 6-min-walk without mask — To walk as fast as possible without running for 6 minutes without mask
  Arms: Without Mask Group

SUMMARY:
Since the beginning of the pandemic caused by SARC-CoV 2, more than 81 million cases have been diagnosed and caused around 1,7 million deaths. Currently, a drug is being sought for the treatment of coronavirus. The worldwide effort to create an effective and safe COVID-19 vaccine is beginning to yield results. Several vaccines now have been authorized around the globe; many more remain in development. Nonetheless, in the absence of effective pharmacological treatment and given the virus's transmission capacity, different alternatives have been proposed to stop the transmission of the virus. Therefore, these preventive measures against transmission are expected to remain in force for some time.

The transmission of the virus occurs from person-to-person; different studies conclude that transmission occurs by aerosols from respiratory droplets. The optimal distance between people to stop person-to-person transmission is uncertain. For this reason and given that there is no effective drug, transmission prevention is of great importance especially for pandemic mitigation in community settings.

The World Health Organization (WHO) established simple precautions to prevent the spread of the virus such as physical distancing, wearing a mask, keeping rooms well ventilated, avoiding crowds, cleaning your hands, and coughing into a bent elbow or tissue. For this reason, the use of the mask has been proposed in several countries, being mandatory in many of them, for use in the health environment and daily use.

The WHO recommends different types of masks depending on the person, where it will be used, or the population incidence in the area. Wearing a medical /surgical mask is recommended for people over 60, those who have underlying medical conditions, feel unwell, and/or look after an ill family member. For health workers, respirator masks (such as FFP2, FFP3, N95, N99) should be used in settings where procedures are generating aerosols.

The use of a mask could imply an inspiratory and expiratory restraint and generate a feeling of discomfort in many people. It is responsible for an increase in the inspiratory and expiratory pressures generated. This feeling of discomfort and the increment of pressures causes shallow and forced breathing and increases the respiratory accessory musculature activation.

Person et al. observed that the subjects who used a mask felt dyspnea clinically and significantly higher than those who did not use it. However, to our knowledge, no study has analyzed the parameters of physical effort, respiratory parameters, self-perceived dyspnea, and muscle activation using different types of masks in healthy subjects. For this reason, the present study hypothesis is that there are no changes between wearing and not-wearing a mask (surgical or N-95) in the effort and ventilatory parameters, even though there may be an increase in the tone of the cervical muscles or the perception of dyspnea using a face mask.

This study aims to observe the effect that the surgical mask and the N-95 mask have in the distance walked, in the oxygenometry, in the heart rate, in the sensation of dyspnea, and the tone of the inspiratory accessory muscles during the 6 minutes walking test.

Procedure After verifying that the subjects meet the inclusion criteria and sign the consent, they will be given a registration number. An investigator will observe the number in a random list and included the participant in one of the three groups (without a mask, with a surgical mask, and with N95 mask). This researcher will make an initial registration of demographic data (gender, age, weight, height, cardiorespiratory pathology, smoker, number of cigarettes per day, a sport performed, hours of daily sport, and days of sport per week). Before the test, all the subjects will have to remain for 30 minutes without a mask, breathing normally. This phase will be called the resting phase. Subsequently, the subjects will go to the area where the 6MWT will be carried out. Each one of them will be performed the test according to the group to which they will be assigned. An investigator, blinded to the subsequent assessment, will encourage the participants to take the 6MWT according to the recommendations mentioned above. After performing the 6MWT, all subjects will go to the assessment area. All the subjects will wear a surgical mask so that the researcher can not know to which group they have been assigned. Besides, this researcher will not have access to the registration number or the 6-minute walking test area.

At the end of each resting phase, SpO2 and baseline HR will be recorded. After every 6MWT, the HR, SpO2, and self-perceived dyspnea will be recorded. The muscle tone will also be assessed with the MyotonPRO in middle scalene and SCM.

Subjects will have the option of retaking the test, going through all the phases mentioned above.

DETAILED DESCRIPTION:
Since the beginning of the pandemic caused by SARC-CoV 2, more than 81 million cases have been diagnosed and caused around 1,7 million deaths. Currently, a drug is being sought for the treatment of coronavirus. The worldwide effort to create an effective and safe COVID-19 vaccine is beginning to yield results. Several vaccines now have been authorized around the globe; many more remain in development. Nonetheless, in the absence of effective pharmacological treatment and given the virus's transmission capacity, different alternatives have been proposed to stop the transmission of the virus. Therefore, these preventive measures against transmission are expected to remain in force for some time.

The transmission of the virus occurs from person-to-person; different studies conclude that transmission occurs by aerosols from respiratory droplets. The optimal distance between people to stop person-to-person transmission is uncertain. For this reason and given that there is no effective drug, transmission prevention is of great importance especially for pandemic mitigation in community settings.

The World Health Organization (WHO) established simple precautions to prevent the spread of the virus such as physical distancing, wearing a mask, keeping rooms well ventilated, avoiding crowds, cleaning your hands, and coughing into a bent elbow or tissue. For this reason, the use of the mask has been proposed in several countries, being mandatory in many of them, for use in the health environment and daily use.

The WHO recommends different types of masks depending on the person, where it will be used, or the population incidence in the area. Wearing a medical /surgical mask is recommended for people over 60, those who have underlying medical conditions, feel unwell, and/or look after an ill family member. For health workers, respirator masks (such as FFP2, FFP3, N95, N99) should be used in settings where procedures are generating aerosols.

The use of a mask could imply an inspiratory and expiratory restraint and generate a feeling of discomfort in many people. It is responsible for an increase in the inspiratory and expiratory pressures generated. This feeling of discomfort and the increment of pressures causes shallow and forced breathing and increases the respiratory accessory musculature activation.

Person et al. observed that the subjects who used a mask felt dyspnea clinically and significantly higher than those who did not use it. However, to our knowledge, no study has analyzed the parameters of physical effort, respiratory parameters, self-perceived dyspnea, and muscle activation using different types of masks in healthy subjects. For this reason, the present study hypothesis is that there are no changes between wearing and not-wearing a mask (surgical or N-95) in the effort and ventilatory parameters, even though there may be an increase in the tone of the cervical muscles or the perception of dyspnea using a face mask.

This study aims to observe the effect that the surgical mask and the N-95 mask have in the distance walked, in the oxygenometry, in the heart rate, in the sensation of dyspnea, and the tone of the inspiratory accessory muscles during the 6 minutes walking test.

Procedure After verifying that the subjects meet the inclusion criteria and sign the consent, they will be given a registration number. An investigator will observe the number in a random list and included the participant in one of the three groups (without a mask, with a surgical mask, and with N95 mask). This researcher will make an initial registration of demographic data (gender, age, weight, height, cardiorespiratory pathology, smoker, number of cigarettes per day, a sport performed, hours of daily sport, and days of sport per week). Before the test, all the subjects will have to remain for 30 minutes without a mask, breathing normally. This phase will be called the resting phase. Subsequently, the subjects will go to the area where the 6MWT will be carried out. Each one of them will be performed the test according to the group to which they will be assigned. An investigator, blinded to the subsequent assessment, will encourage the participants to take the 6MWT according to the recommendations mentioned above. After performing the 6MWT, all subjects will go to the assessment area. All the subjects will wear a surgical mask so that the researcher can not know to which group they have been assigned. Besides, this researcher will not have access to the registration number or the 6-minute walking test area.

At the end of each resting phase, SpO2 and baseline HR will be recorded. After every 6MWT, the HR, SpO2, and self-perceived dyspnea will be recorded. The muscle tone will also be assessed with the MyotonPRO in middle scalene and SCM.

Subjects will have the option of retaking the test, going through all the phases mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Being able to perform the 6 min-walk-test-

Exclusion Criteria:

* Cardiac-respiratory diseases
* Red flags.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-10 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
6 minutes walk test (minutes) | Change between baseline (immediately before intervention) and post intervention (immediately after intervention)
  The volunteers had to walk as fast as possible without running for 6 minutes. Each minute, the subjects will be encouraged to continue at the same pace and not stop

SECONDARY OUTCOMES:
Dyspnea using the visual analogue scale (VAS) (cms) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  Dyspnea sensation in the visual analogue scale (0 to 100 cms).
Heart Rate (b/min) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  With a pulse oximeter (b/min).
Transcutaneous oxygen saturation (% of saturation) | Change between baseline(immediately before intervention) and post intervention (immediately after intervention)
  With a pulse oximeter (SpO2).
Frequency Muscle tone with MyotonePRO device (Hz) | Change between baseline and post intervention (1 month), after 3 months and after 6 months
  The Myoton PRO device will be used to register the respiratory accessory muscle tone. This handheld device was designed to assess the muscle and its characteristics. A brief mechanical impulse on the skin generates a natural oscillation of the tissues that cushion it.
Dynamic Stiffness Muscle tone with MyotonePRO device (N/m) | Change between baseline and post intervention (1 month), after 3 months and after 6 months
  The Myoton PRO device will be used to register the respiratory accessory muscle tone. This handheld device was designed to assess the muscle and its characteristics. A brief mechanical impulse on the skin generates a natural oscillation of the tissues that cushion it.
Muscle viscoelasticy with MyotonePRO device (ms) | Change between baseline and post intervention (1 month), after 3 months and after 6 months
  The Myoton PRO device will be used to register the respiratory accessory muscle tone. This handheld device was designed to assess the muscle and its characteristics. A brief mechanical impulse on the skin generates a natural oscillation of the tissues that cushion it.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Pérez-Bellmunt, PhD, Study Director — Universitat Internacional de Catalunya
Locations (2):
- Spain (2):
  - Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona
  - Universitat Internacional de Catalunya, Sant Cugat del Vallès

IPD SHARING:
Plan to Share IPD: No